CLINICAL TRIAL: NCT01853709
Title: Multidisciplinary Approach Versus Conventional Approach in Colonic Preparation of Hospitalized Patients. A Randomized Controlled Trial
Brief Title: Multidisciplinary Approach Versus Conventional Approach in Colonic Preparation of Hospitalized Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Felix Junquera, Consultant Physician - Gastroenterology, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPT-END-DIG-2012
Record Dates: First submitted 2013-04-29; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Bowel Preparation for Colonoscopy
MeSH Terms: interventions — Educational Status; Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary approach (Experimental): The multidisciplinary approach will include:
  Education Fiber free diet Bisacodyl: 10 mg 2 days before the procedure, 20 mg the day before the procedure and 10 mg 3 hours before the procedure Adjuvants: Olive Oil:60 mL/Apple Juice: 200 mL PEG: 1 L the night before the procedure and 1 L 3 hours before the procedure
  Interventions: Behavioral: Education; Other: Fiber free diet; Dietary Supplement: Adjuvants; Drug: Polyethylene glycol (PEG); Drug: Bisacodyl
- Conventional approach (Active Comparator): The conventional approach will include:
  Education Fiber free diet Polyethylene glycol (PEG): 2 L the night before the procedure, 2 L 3 hours before the procedure
  Interventions: Behavioral: Education; Other: Fiber free diet; Drug: Polyethylene glycol (PEG)

INTERVENTIONS:
Behavioral: Education
Other: Fiber free diet
Dietary Supplement: Adjuvants
  Arms: Multidisciplinary approach
Drug: Polyethylene glycol (PEG)
Drug: Bisacodyl
  Arms: Multidisciplinary approach

SUMMARY:
Colonoscopy is the gold standard diagnostic procedure for colonic disease. Excellent bowel cleansing is critical for this procedure. However, an inadequate bowel cleansing is a common problem that occurs up to 20% of procedures. This fact has a deep clinical and economical impact. In fact, inadequate bowel preparation is associated to misdiagnosis in 30% of lesions. Moreover several clinical conditions such as cirrhosis, antidepressant drugs, and hospitalized patients are predictive factors of inadequate colonic preparations. These circumstances have promoted multiple clinical trials, however there is no consensus about the optimal strategy for colonic cleansing. Education in colonic preparation has obtained conflicting results. Polyethylene glycol (PEG) and sodium phosphate solutions have been the commonest preparations used with a similar efficacy. However, the large volume to ingest (4 litters) makes PEG compliance difficult. Likewise, sodium phosphate also contains high levels in sodium and phosphate which contraindicate its use in elderly patients and / or with comorbidity. The use of adjuvants such as olive oil and bisacodyl allows reducing the volume of polyethylene glycol thereby improving the tolerance and right colon preparation.

The aim of this study is to compare the efficacy of a multidisciplinary approach (education, fiber free diet, polyethylene glycol (PEG) 2L, and adjuvant bisacodyl + olive oil) vs. a conventional approach (fiber free diet+ PEG 4L in split doses ) in cleaning the colon of hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who undergo a non urgent colonoscopy
* Patients who give informed consent to participate in the study
* Patients older than 18 years
* Patients who undergo total colonoscopy

Exclusion Criteria:

* Non compliance with the 48 hours diet prescribed
* The endoscopy planned is a rectosigmoidoscopy
* Previous colonic surgery
* Mental/cognitive impairment preventing the study assessments
* Severe renal failure
* Electrolytic disbalance(hyponatremia, hypokaliemia, Hyperphosphatemia, hypocalcemia and hypomagnesemia)
* Intestinal obstruction, perforation or toxic megacolon
* Pregnant or nursing women
* Allergy/intolerance to PEG, bisacodyl or adjuvants
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with adequate bowel preparation | at the time of performing the colonoscopy
  Adequate bowel preparation is defined as a preparation which allows exploring the whole colonic mucose and detecting flat lesions (Rating as good or excellent in the Boston Bowel preparation scale)

SECONDARY OUTCOMES:
Percentage of patients with adequate bowel preparation by bowel segments | At the time of performing the colonoscopy
  The boston scale will be assessed by the investigators during the procedure.
Tolerance to the colonoscopy | from colonoscopy up to 24 hours after colonoscopy
  Tolerance to the colonoscopy will be measured by VAS during the colonoscopy, 30 minutes after colonoscopy and 24 hours after colonoscopy
Percentage of complete/incomplete colonoscopies and reprogramming | After the colonoscopy
  Evaluation of incomplete or inadequate bowel preparation will be assessed after performing the colonoscopy
Complications during and after the procedure | up to 24 hours after colonoscopy
Doses of sedation needed during the colonoscopy | During the colonoscopy process
  Final dose will be calculated at the end of the procedure
Tolerance to the preparation | up to 48 hours
Endoscopic findings | during the colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain